CLINICAL TRIAL: NCT03194607
Title: Quantitative Evaluation of Motor Function Before and After Surgery for Degenerative Lumbar Spinal Stenosis
Acronym: SPEED
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GRELAT 2016
Record Dates: First submitted 2017-06-15; First posted 2017-06-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Posture; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Patients
  Interventions: Other: Functional walk tests; Other: 3D analysis of locomotion and posture; Other: questionnaires
- Controls
  Interventions: Other: Functional walk tests; Other: 3D analysis of locomotion and posture; Other: questionnaires

INTERVENTIONS:
Other: Functional walk tests
Other: 3D analysis of locomotion and posture
Other: questionnaires

SUMMARY:
Low back pain is a leading cause of medical consultations in France and in other industrialized countries. Although spinal surgery is a recognized treatment, to date, its impact has only been assessed using subjective or declarative criteria. Yet, in many orthopaedic diseases, it has been shown that the evaluation of functional capacities, including walking speed, is particularly useful to study the impact of these diseases and their treatment. To date, no study has attempted to assess the impact of spinal surgery by evaluating 1) the functional capacities of patients and 2) spatio-temporal parameters of locomotion and joint dynamics. The investigators hypothesize that spinal surgery in patients with symptomatic lumbar spinal stenosis should lead to an improvement in quantifiable locomotion parameters, and in particular walking speed. Walking speed is a quantitative measurement, which could reflect the degree of functional impairment of the patient before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

Patient:

* more than 18 years old
* who has provided verbal consent
* with acquired arthritic lumbar spinal stenosis
* eligible for surgery (pain > 3 months, resistant to medical treatment)
* for whom the neurosurgeon has scheduled nerve decompression without osteosynthesis or instrumentation
* able to walk ≥ 10 metres without help

Exclusion Criteria:

Patient:

* Adult under guardianship
* Absence of health insurance cover
* Pregnant or breast-feeding women
* History of lumbar spinal surgery involving posterior or anterior arthrodesis
* History of lumbar spinal surgery involving arthroplasty
* History of lumbar spinal surgery within the previous 12 months
* Locomotor disorders due to causes other than spine disease (orthopaedic, neurological, vascular, cardiac…) that could significantly affect walking speed
* patients in whom the surgery could not be done or deferred (intolerance to the ventral decubitus position, infection…)
* patients who had revisit surgery before M6 (with the exception of early revisit surgery during the first month post-intervention)
* patients in whom osteosynthesis or the implantation of instruments was decided and done during the surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: low back pain lumbar spinal stenosis spinal surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Compare the free walking speed in patients (6-minute walk test), before and after surgery | 2 weeks and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Gouteron A, Laroche D, Beaurain J, Ksiazek E, Fournel I, Bohm A, Ornetti P, Casillas JM, Armand S, Gueugnon M. Effect of decompression surgery for lumbar spinal stenosis on aerobic capacities during a 6-min walk test: A preliminary cohort study. Ann Phys Rehabil Med. 2023 Mar;66(2):101673. doi: 10.1016/j.rehab.2022.101673. Epub 2022 Dec 1. No abstract available. PMID 35489687
- [Derived] Gueugnon M, Riglet L, Fournel I, Ksiazek E, Beaurain J, Chapon R, Ornetti P, Laroche D. Evaluation of the sagittal vertical axis with postural and 3D motion analyses in lumbar spinal stenosis. BMC Musculoskelet Disord. 2024 Oct 19;25(1):827. doi: 10.1186/s12891-024-07923-y. PMID 39427140